CLINICAL TRIAL: NCT00779610
Title: The Effects of Passive and Active Vibration Therapy on Grip Strength and Myoelectric Activity
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. John Zhang, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR0810080147
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Strength
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Vibration with forearm flexion (active contraction)
  Interventions: Procedure: Vibration with flexion
- Passive (Sham Comparator): Vibration without forearm flexion (passive)
  Interventions: Procedure: Vibration without flexion

INTERVENTIONS:
Procedure: Vibration with flexion — Vibration with forearm flexion (active contraction)
  Arms: Active
Procedure: Vibration without flexion — Vibration without forearm flexion (passive)
  Arms: Passive

SUMMARY:
This pilot study is designed to analyze the effects of Vibration Therapy (VT) on grip strength and level of forearm contraction by measuring hand grip dynamometry and surface Electromyography (sEMG) using the BioPac sEMG and digital dynamometry devices after the application of both passive and active Vibrational Therapy (VT) using the PowerPlate.

ELIGIBILITY:
Inclusion Criteria:

* participants will be Logan students, faculty and staff 18-65 yoa
* asymptomatic subject will be included in the study
* participants must complete a survey and consent form
* only participants that meet the criteria of the survey will be accepted in the study

Exclusion Criteria:

* participant with any recent or past disease/injuries/trauma/fracture (i.e., arthritis, carpal tunnel, etc.)
* who have had joint replacements
* who are currently engaging in physical rehabilitation
* who are pregnant will be excluded from the study
* history of cardiovascular disease
* history of cancer
* history of epilepsy
* history of diabetes mellitus, or past retinal surgeries
* participants cannot have Chiropractic manipulation or engage in weight lifting or other extreme exercise throughout the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Surface EMG and Grip Strength Dynamometry | Pre and Post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States